CLINICAL TRIAL: NCT00583128
Title: A Double-Blind, Randomized, Placebo-Controlled Multicenter Study to Assess the Safety and Efficacy of AST-120 in Patients With Non-Constipating Irritable Bowel Syndrome
Brief Title: Safety and Efficacy of AST-120 in Patients With Non-Constipating Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ocera Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AST014
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — AST 120

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AST-120, 2 gram sachets
  Interventions: Drug: AST-120
- 2 (Placebo Comparator): Celphere® CP-305, stained to match appearance of AST-120, in 2g sachets
  Interventions: Drug: Celphere® CP-305

INTERVENTIONS:
Drug: AST-120 — oral, sachet, 2 grams three times daily for 8 weeks
  Arms: 1
Drug: Celphere® CP-305 — oral, placebo, sachet, 2 grams three times daily for 8 weeks
  Arms: 2

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the experimental drug AST-120 in treating patients with non-constipating IBS. The study will test whether or not patients receiving AST-120 experience at least a 50% reduction in the number of days with abdominal pain compared to placebo.

DETAILED DESCRIPTION:
Patients experiencing non-constipating IBS will be randomized to one of two arms in the study: the experimental drug AST-120 or placebo. Patients will take 2g of AST-120 or placebo three times per day for eight weeks. After the 8 week course, patients will receive an additional 8 weeks single blind treatment, after a one week washout period.

The experimental drug AST-120 is composed of black, odorless spherical carbon particles in 2g sachets (aluminum foil pouches). The placebo consists of microcrystalline cellulose spheres, Celphere CP-305 stained to match the appearance of AST-120, in 2g sachets (aluminum foil pouches). Both AST-120 and placebo are oral (taken by mouth) preparations. Both are tasteless. To take the product, patients will tear open the sachet, drop the contents directly on their tongue and wash it down with 8 ounces of water.

Patients will be expected to participate in up to 10 visits, approximately three by telephone and the remainder of visits are in-clinic. At these visits, patients will undergo a number of tests including: hematology panel, lactose intolerance testing, physical exams, pregnancy tests, evaluations based on the following scales: The Bristol Stool Scale, IBS Severity Scale, IBS Quality of Life, SCL-90R.

Provided the patient has been stable for eight weeks prior to their baseline visit, they will be allowed to take the following medications: drugs that inhibit gastric secretion (histamine blockers, proton pump inhibitors), benzodiazepines and Imidazopyridines (short acting, nonbenzodiazepine hypnotics) for sleep (dose must be consistent with the use of a sleep agent) aspirin at a cardiovascular prophylactic dose (75-150 mg/day) and paracetamol. Antidepressants for non-IBS symptoms are allowed. Loperamide will be permitted as a rescue for diarrhea only when patients are experiencing at least 3 liquid or soft stools in one day. However, Loperamide is prohibited during the two week screening period.

Patients will not be allowed to take the following medications whilst on trial and these therapies must have been discontinued by at least two weeks prior to their baseline visit: probiotics, neuroleptics, antidepressants for IBS symptoms, daytime tranquilizers, prokinetics, spasmolytics, analgesics, other investigational agents and any over-the-counter medications.

Patient will be required to keep a diary during the study

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥ 40 kg;
* Recurrent abdominal pain or discomfort for three or more days per month for the last three months which meets Rome III criteria for non-constipating IBS;
* Patients on a stable diet for at least eight weeks;
* Patients ≥ 50 years of age with a negative screening colonoscopy in the last five years;
* Able and willing to comply with all protocol procedures for the planned duration of the study;
* Able and willing to understand, sign and date an informed consent document, and authorize access to protected health information,
* Females must be postmenopausal, surgically incapable of bearing children, or practicing a reliable method of birth control (intrauterine devices, spermicide and barrier) (Hormonal contraceptives are NOT regarded as adequate for the purpose of this trial.) Partner/spouse sterility may also qualify at the Investigator's discretion. Females of child-bearing potential must have a negative urine pregnancy test at baseline.

Exclusion Criteria:

* Constipating IBS;
* History of untreated lactose intolerance;
* History of colonic or major abdominal surgery (colectomy, for example);
* Active (untreated) Thyroid disease;
* Current diagnosis of major depression or psychosis;
* Known positive stool cultures for Clostridium difficile or other pathogens;
* Any condition necessitating the administration of analgesics (except paracetamol), probiotics, neuroleptics, antidepressants for IBS symptoms, daytime tranquilizers, prokinetics or spasmolytic medications;
* Poor tolerability of venipuncture or lack of adequate venous access for required blood sampling;
* Other major physical or major psychiatric illness within the last six months that in the opinion of the investigator would affect the patient's ability to complete the trial;
* Uncontrolled systemic disease such as diabetes;
* Patients undergoing chemotherapy for the treatment of cancer;
* Known hypersensitivity or contraindication to any component of the test product (study drugs) or diagnostics used;
* Participation in another study within eight (8) weeks prior to the study;
* Unable to attend all visits required by the protocol;
* Female patients must be excluded if they are pregnant, breast feeding, or planning to become pregnant during the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2007-08; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Percent of patients who achieve at least a 50% reduction in the number of days with abdominal pain during the final 2 weeks of the double-blind treatment course. | Eight weeks
Safety endpoint is adverse events (AEs) deemed possibly, probably, or definitely related to treatment with investigational product during the double-blind treatment course. | 8 weeks

SECONDARY OUTCOMES:
Percent change in the IBS QOL score. | Eight weeks
Percent change in HADS score. | 8 weeks
Percent change in Bristol Scale score. | 8 weeks
Percent change in individual items in the IBS Symptom Severity questionnaire. | 8 weeks
Durability of effect after the first eight weeks of treatment. | 8 weeks
Change in clinical laboratory tests from Baseline to Week 8 and to Week 18. | 8 weeks
Any adverse event occurring after Week 8. | 8 weeks
Physical examinations, vital signs (blood pressure, heart rate, respiration and temperature). | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, MD, Principal Investigator — University of Leuven, Department of Gastroenterology
Locations (17):
- United States (13):
  - Clinical Research Associates, Huntsville, Alabama
  - Northern California Research, Sacramento, California
  - Medical Center for Clinical Research, San Diego, California
  - Madeleine DuPree, MD, Boynton Beach, Florida
  - Michael Epstein, MD, Annapolis, Maryland
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Long Island Gastrointestinal Research Group, Great Neck, New York
  - LeBauer Research Associates, Greensboro, North Carolina
  - Peters Medical Research, LLC, High Point, North Carolina
  - Ohio Gastroenterology and Liver Institute, Cincinnatti, Ohio
  - Oklahoma Foundation for Digestive Disease, Oklahoma City, Oklahoma
  - Breco Research LTD, Houston, Texas
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin
- Belgium (4):
  - Zuid-Oost Limburg Campus St. Jan, Genk, Genk
  - UCL St. Luc, Woluwe, Woluwe
  - AZ St. Lucas Assebroek, Assebroek
  - UZ Leuven, Leuven

REFERENCES:
- [Background] Drossman DA. The functional gastrointestinal disorders and the Rome III process. Gastroenterology. 2006 Apr;130(5):1377-90. doi: 10.1053/j.gastro.2006.03.008. No abstract available. PMID 16678553
- [Background] Schuster MM. Defining and diagnosing irritable bowel syndrome. Am J Manag Care. 2001 Jul;7(8 Suppl):S246-51. PMID 11474909
- [Background] Tack J, Broekaert D, Fischler B, Van Oudenhove L, Gevers AM, Janssens J. A controlled crossover study of the selective serotonin reuptake inhibitor citalopram in irritable bowel syndrome. Gut. 2006 Aug;55(8):1095-103. doi: 10.1136/gut.2005.077503. Epub 2006 Jan 9. PMID 16401691
- [Background] Wood JD. Histamine, mast cells, and the enteric nervous system in the irritable bowel syndrome, enteritis, and food allergies. Gut. 2006 Apr;55(4):445-7. doi: 10.1136/gut.2005.079046. PMID 16531524
- [Result] Tack JF, Miner PB Jr, Fischer L, Harris MS. Randomised clinical trial: the safety and efficacy of AST-120 in non-constipating irritable bowel syndrome - a double-blind, placebo-controlled study. Aliment Pharmacol Ther. 2011 Oct;34(8):868-77. doi: 10.1111/j.1365-2036.2011.04818.x. Epub 2011 Aug 24. PMID 21883322